CLINICAL TRIAL: NCT02916355
Title: Role of IL-1 in Postprandial Fatigue - The Chäschüechli 2 Study
Brief Title: Role of Interleukin (IL)-1 in Postprandial Fatigue - The Chäschüechli 2 Study
Acronym: Chäs2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: EKNZ BASEC 2016-00816
Record Dates: First submitted 2016-09-26; First posted 2016-09-27 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Adiposity
MeSH Terms: conditions — Obesity | interventions — Interleukin 1 Receptor Antagonist Protein; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal BMI (Experimental): Healthy young men, normal BMI (BMI >18 and ≤28 kg/m2) will receive interventions Anakinra and sodium Chloride (NaCl)
  Interventions: Drug: Anakinra; Drug: NaCl
- Overweight (Experimental): Healthy young men (BMI >30 and ≤35 kg/m2) will receive interventions Anakinra and NaCl
  Interventions: Drug: Anakinra; Drug: NaCl

INTERVENTIONS:
Drug: Anakinra — Subjects will receive Anakinra infusion and afterwards they will be fed a very fat containing meal, and postprandial fatigue will be measured regularly until 3,5 hour after the meal.
  Other Names: Kineret
Drug: NaCl — subjects will receive NaCl infusion and afterwards they will be fed a very fat containing meal, and postprandial fatigue will be measured regularly until 3,5 hour after the meal.
  Other Names: sodium chloride

SUMMARY:
Role of IL-1 in postprandial fatigue - The Chäschüechli 2 Study It is a randomized, single dose, placebo-controlled, double blind, cross-over, proof-of-concept study.

16 healthy young men will be included in this study. The objective of this study is to evaluate if severity of postprandial fatigue is driven by IL-1.

Since fatigue is associated with increased cytokine levels, and since fatigue in chronic inflammatory settings, such as type 2 diabetes, can be reduced by inhibition of IL-1β, postprandial fatigue might also respond to anti-inflammatory intervention with IL-1 inhibition.

The aim of the study is to investigate whether postprandial fatigue is, at least in part, driven by the IL-1 system.

ELIGIBILITY:
Inclusion Criteria:

Male subjects

* non-smoking
* apparently healthy
* BMI >18 and ≤28 kg/m2 or BMI >30 and ≤35 kg/m2
* Age 20-65 years
* Subject is usually eating breakfast and lunch
* Willingness to use contraceptive measures adequate to prevent the subject's partner from becoming pregnant during the study. Adequate contraceptive measures include hormonal methods used for two or more cycles prior to screening (e.g., oral contraceptive pills, contraceptive patch, or contraceptive vaginal ring), double barrier methods (e.g., contraceptive sponge, diaphragm used in conjunction with contraceptive foam or jelly, and condom used in conjunction with contraceptive foam or jelly), intrauterine methods (IUD) and sterilization (e.g., tubal ligation or a monogamous relationship with a vasectomized partner).
* Owner of a smartphone so they will be able to download and use the sleeping APP, Sleep cycle, prior to the study days.

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the following criteria:

* Night shift workers
* Subjects suffering from sleep disturbances
* Clinical signs of infection in the week before inclusion or history of infection during the last 2 months (CRP >5mg/l)
* Impaired fasting glucose (fasting plasma glucose >5.5mmol/l)
* Hematologic disease (leukocyte count < 1.5x109/l, hemoglobin <11 g/dl, platelets <100 x 103/ul)
* Kidney disease (creatinine > 1.5 mg/dl))
* Liver disease (transaminases >2x upper normal range)
* Heart disease
* Pulmonary disease
* Inflammatory disease
* History of carcinoma
* History of tuberculosis
* Alcohol consumption >40g/d
* Smoking
* Known allergy towards Kineret
* Known allergy to ingredients of the test meal
* Current treatment with any drug in the week before inclusion, including vitamin supplementation (especially vitamin C and E)
* Use of any investigational drug within 30 days prior to enrolment or within 5 half-lives of the investigational drug, whichever is longer
* Subject refusing or unable to give written informed consent

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-08; Primary Completion 2017-04 (Actual); Study Completion 2017-04-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome is change in fatigue measured by the SSS (Stanford Sleepiness Scale) between groups treated with Anakinra vs. placebo | 7 to 9 days (change between study day 1 and study day 2)
  Fatigue will be measured by using the SSS (Stanford Sleepiness Scale)

SECONDARY OUTCOMES:
Change in postprandial glucose, insulin, C-peptide, glucagon-like Peptide (GLP)-1(active/total), GIP(active/total), PYY, IL-6, tumor necrosis factor (TNF)-alfa, sCRP and cortisol due to any treatment (Anakinra vs. saline). | 7 to 9 days (change between study day 1 and study day 2)
  Blood sampling
Change in heart rate due to any treatment (Anakinra vs. saline) | 7 to 9 days (change between study day 1 and study day 2)
  Pulse watch
Change in insulin due to any treatment (Anakinra vs. saline). | 7 to 9 days (change between study day 1 and study day 2)
  Blood sampling
Change in C-peptide due to any treatment (Anakinra vs. saline). | 7 to 9 days (change between study day 1 and study day 2)
  Blood sampling
Change in GLP-1(active/total) due to any treatment (Anakinra vs. saline). | 7 to 9 days (change between study day 1 and study day 2)
  Blood sampling
Change in GIP(active/total) due to any treatment (Anakinra vs. saline). | 7 to 9 days (change between study day 1 and study day 2)
  Blood sampling
Change in PYY due to any treatment (Anakinra vs. saline). | 7 to 9 days (change between study day 1 and study day 2)
  Blood sampling
Change in IL-6 due to any treatment (Anakinra vs. saline). | 7 to 9 days (change between study day 1 and study day 2)
  Blood sampling
Change in TNF-alfa due to any treatment (Anakinra vs. saline). | 7 to 9 days (change between study day 1 and study day 2)
  Blood sampling
Change in sCRP due to any treatment (Anakinra vs. saline). | 7 to 9 days (change between study day 1 and study day 2)
  Blood sampling
Change in cortisol due to any treatment (Anakinra vs. saline). | 7 to 9 days (change between study day 1 and study day 2)
  Blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Marc Y Donath, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Department of Endocrinology, Diabetes and Metabolism, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No